CLINICAL TRIAL: NCT02955836
Title: Establishing and Exploring the Need and Effectiveness of Monitoring Information System of Nursing-related Patient Safety and Quality Indicators
Brief Title: Effectiveness of Monitoring Information System of Nursing Related Patient Safety and Quality Indicators
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201610021RINB
Record Dates: First submitted 2016-10-31; First posted 2016-11-04 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-11

CONDITIONS: Patient Safety; Quality Indicator; Information System; Nursing; Healthcare Quality
Keywords: Patient Safety; Quality indicator; Information system; Nursing; Healthcare Quality; Quality measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: The purposes of this study are 1) to understand the nurses' need and perception toward of the monitoring information system of nursing-related patient safety and quality indicators; 2) to establish the monitoring information system of nursing-related patient safety and quality indicators; 3) to evaluate the monitoring information system of nursing-related patient safety and quality indicators.

Methods: There will be three phases and the study site in the medical center in northern Taiwan. The first phase is information needs assessment. Researchers will hold the meeting of focus group discussion. The subjects will be the nursing manager, head nurse, clinical nurses who are similar to nursing-related patient safety and quality indicators. The self-conducted semi-structure discussion form will be used to collect the data during the meeting of focus group discussion. The questionnaire will be used to collect the perception, attitude, behavior, satisfaction, time-consuming and the accuracy of nursing-related patient safety and quality indicators data from nurses. The second phase will establish the monitoring information system of nursing-related patient safety and quality indicators and clinical implementation. The third phase will evaluate the effectiveness of the monitoring information system of nursing-related patient safety and quality indicators. The questionnaire will be used to collect the satisfaction, time-consuming and the accuracy of nursing-related patient safety and quality indicators from nurses during the evaluation phase.

DETAILED DESCRIPTION:
Background: Monitoring the patient safety and quality of nursing care is essential to identify patients at risk. Monitoring the nursing-related patient safety and quality indicators are important for high-quality nursing care. However, monitoring nursing-related patient safety and quality indicators through information system is a challenge. The nurses' to date workload is increasing. The comprehensive nursing-related patient safety and quality indicators information system should be used to make nurses work of collecting indicator data more efficiency and enhance patient care quality.

Objective: The purposes of this study are 1) to understand the nurses' need and perception toward of the monitoring information system of nursing-related patient safety and quality indicators; 2) to establish the monitoring information system of nursing-related patient safety and quality indicators; 3) to evaluate the monitoring information system of nursing-related patient safety and quality indicators.

Methods: There will be three phases and the study site in the medical center in northern Taiwan. The first phase is information needs assessment. Researchers will hold the meeting of focus group discussion. The subjects will be the nursing manager, head nurse, clinical nurses who are similar to nursing-related patient safety and quality indicators. The self-conducted semi-structure discussion form will be used to collect the data during the meeting of focus group discussion. The questionnaire will be used to collect the perception, attitude, behavior, satisfaction, time-consuming and the accuracy of nursing-related patient safety and quality indicators data from nurses. The second phase will establish the monitoring information system of nursing-related patient safety and quality indicators and clinical implementation. The third phase will evaluate the effectiveness of the monitoring information system of nursing-related patient safety and quality indicators. The questionnaire will be used to collect the satisfaction, time-consuming and the accuracy of nursing-related patient safety and quality indicators from nurses during the evaluation phase.

Expected results: The investigators will understand the nurses' need and perception toward of the monitoring information system of nursing-related patient safety and quality indicators and establish it. After establishing the monitoring information system of nursing-related patient safety and quality indicators, the investigators can obtain the result through information technology to achieve the accuracy of indicator data and the high efficiency of nursing quality control. Moreover, it can decrease the time consuming and burden to collect data of indicators, improve the nurses' and nurse managers' satisfaction and positive experiences. In addition to that, the investigators can also get the goal of creating patient safety and high-quality nursing care.

ELIGIBILITY:
inclusion criteria:

* Registered nurse.

exclusion criteria:

* Registered nurse who are not interested in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: nursing manager, head nurse, clinical nurses
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
satisfaction survey | 2016-2019

SECONDARY OUTCOMES:
survey of time consumption | 2016-2019
survey of the perception, attitude and behavior of quality eMeasures | 2016-2019

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Lien Lin, PhD, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No